CLINICAL TRIAL: NCT00353028
Title: SME3110 (Fluvoxamine Maleate) in the Treatment of Depression/Depressive State : A Post-marketing Clinical Study in Children and Adolescents (8 Through 18 Years of Age) -A Double-blind, Randomized, Placeb-controlled Study
Brief Title: Fluvoxamine Maleate in the Treatment of Depression/Depressive State : A Post-marketing Clinical Study in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S114.3.117
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Major Depressive Disorder
Keywords: Fluvoxamine Maleate; Depression; Children and Adolescents
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- F (Experimental)
  Interventions: Drug: Fluvoxamine maleate
- P (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine maleate — Test product: Fluvoxamine maleate 25mg tablet. In case that the daily dose is one tablet, the study medication will orally be administered once daily, at bedtime. In case that the daily dose is two tablets or higher (maximam:6 tablets), the study mmedica
  Arms: F
Drug: Placebo — Placebo
  Arms: P

SUMMARY:
This study is to verify the efficacy of fluvoxamine maleate given for 8 weeks in the treatment of children and adolescents with depression or depressive state

ELIGIBILITY:
Inclusion Criteria Have a minimum total score of 18 on the JSIGH-D, Weight is within the standard weight ± 2S.D. based on the standard weight for each age in the School Health Statistical Survey Exclusion Criteria Have the following predominant psychiatric diagnosis -Schizophrenia Have previously been treated with fluvoxamine maleate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
the time of onset of 50% decrease from baseline in the Japanese Version of the Structured Interview Guide for the Hamilton Depression Rating Scale (JSIGH-D) 17-item total score | 8 weeks

SECONDARY OUTCOMES:
The Clinical Global Impression(CGI) improvement at Week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Yamaguchi, Study Director — Solvay Pharmaceuticals
Locations (25):
- Japan (25):
  - S114.3.117 Kohnodai Hospital, National Center of N, Chiba Prefecture
  - S114.3.117 Fukuoka University Hospital, Fukuoka Prefecture
  - S114.3.117 Hatakeyama Clinic, Fukuoka Prefecture
  - S114.3.117 Kaname Clinic, Fukuoka Prefecture
  - S114.3.117 Kashi shinryo Clinic, Fukuoka Prefecture
  - S114.3.117 Kashii Sanatorium, Fukuoka Prefecture
  - S114.3.117 Kyushu University Hospital, Fukuoka Prefecture
  - S114.3.117 Shiranui Hospital, Fukuoka Prefecture
  - S114.3.117 Sugahara Tenjin Hospital, Fukuoka Prefecture
  - S114.3.117 Hiroshima-city Funairi Hospital, Hiroshima Prefecture
  - S114.3.117 Goryokai Hospital, Hokkaido Prefecture
  - S114.3.117 Kobe University Hospital, Hyogo Prefecture
  - S114.3.117 National Hospital Organization Kagawa C, Kagawa Prefecture
  - S114.3.117 Yokohama City University Hospital, Kanagawa Prefecture
  - S114.3.117 National Hospital Organization Kikuti N, Kumamoto Prefecture
  - S114.3.117 Kyoto University Hospital, Kyoto Prefecture
  - S114.3.117 National Hospital Organization Sakakiba, Mie Prefecuture
  - S114.3.117 Shinshu University Hospital, Nagano Prefecture
  - S114.3.117 Aichi Children's Health and Medical Cen, Nagoya Prefecture
  - S114.3.117 Nagoya Mental Clinic, Nagoya Prefecture
  - S114.3.117 Nara Medical University Hospital, Nara Prefecture
  - S114.3.117 Kansai Medical University Takii Hospita, Osaka Prefecture
  - S114.3.117 Kusube Clinic, Osaka Prefecture
  - S114.3.117 Yasuhara Children's Clinic, Osaka Prefecture
  - S114.3.117 Tokushima University Hospital, Tokushima Prefecture